CLINICAL TRIAL: NCT01198990
Title: SCALE: Small Changes and Lasting Effects
Acronym: SCALE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Mary E. Charlson, MD, Principal Investigator, Weill Medical College of Cornell University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 0908010566
Record Dates: First submitted 2010-09-08; First posted 2010-09-10 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Eating

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Subjects in will be randomized to the small change eating strategy, a physical activity goal and will receive the positive affect/self affirmation component.
  eating/physical activity/positive affect/self-affirmation group.
  Interventions: Behavioral: Group 1
- Group 2 (Experimental): Subjects will be randomized to the small change eating strategy and a physical activity goal.
  eating/physical activity group. No intervention, just the eating strategy and physical activity components.
  Interventions: Behavioral: Group 2

INTERVENTIONS:
Behavioral: Group 1 — Subjects will be randomized to the small change eating strategy, a physical activity goal and will receive the positive affect/self affirmation component.
  Other Names: eating/physical activity/positive affect/self-affirmation
  Arms: Group 1
Behavioral: Group 2 — Subjects will be randomized to the small change eating strategy and a physical activity goal.
  Other Names: eating strategy and physical activity goal
  Arms: Group 2

SUMMARY:
The goal of this study is to translate basic behavioral and social science discoveries into effective behavioral interventions that reduce obesity and obesity related morbidity in Black and Latino communities. This intervention will focus on promoting small changes in eating behavior and increasing physical activity among Black and Latino participants in Harlem and the South Bronx. The desired result from these activities is individual weight loss that will be sustained years after participation in the study.

DETAILED DESCRIPTION:
SCALE is a five year study (October 1, 2009 through June 30, 2014) funded by NHLBI. The study will examine the possibility and acceptance of a mindful eating intervention in African American and Latino participants. We will test whether positive thinking can protect participants against the negative impact that stress and depression can have on making positive behavior changes such as mindful eating and physical activity.

Currently, the SCALE study is in the trial phase. Among overweight or obese Black or Latino adults who live in Harlem or the South Bronx, the primary goal of this project is to achieve weight loss of 7% or more over 12 months by making small sustained changes in eating behavior coupled with sustained increases in physical activity. Participants are enrolled for 12 months and are randomized to one of two study groups.

Group 1: Will choose one of ten small change eating strategies, a physical activity goal and will receive the positive affect/self affirmation component.

Group 2: Will choose one of ten small change eating strategies and a physical activity goal

For inquiries regarding potential enrollment in this study, please contact Rosio Ramos at 646-962-5070 or email ror2023@med.cornell.edu

ELIGIBILITY:
Inclusion Criteria:

Eligibility Criteria:

Black or Latino community-dwelling subjects who are 21 years or older and have a body mass index of >25 but <50 or considered to be obese or overweight are be eligible for study participation. All participants must be able to participate in physical activity and Must be fluent in English or Spanish.

Exclusion Criteria:

Subjects will be excluded if:

1. Unable to provide informed consent in either English or Spanish for any reason, including cognitive impairment, psychiatric illness, drug or alcohol addiction
2. Pregnant or are planning to become pregnant within the year
3. Participating in another weight loss program or trial
4. On medications for obesity
5. Have a history of bulimia;
6. history of surgery for obesity;
7. Have severe comorbid diseases that can lead to unintentional weight change including cancer, HIV/AIDS, congestive heart failure.
8. They live in an institutional setting (nursing home, prison or group home).
9. Have severe disease or are terminally ill, including stroke, myocardial infarction, coronary artery disease requiring angioplasty.

   -

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2009-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Percent weight loss | 12 months
  The primary goal of this project is to achieve weight loss of 7% or more over 12 months by making small sustained changes in eating behavior coupled with sustained increases in physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Charlson, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (6):
- United States (6):
  - Renaissance Health Care Network, New York, New York
  - Abyssinian Baptist Church, New York, New York
  - Metropolitan Methodist Church, New York, New York
  - Lincoln Medical and Mental Health Center, The Bronx, New York
  - East Side House Settlement, The Bronx, New York
  - Iglesia Congregacion Cristiana del Bronx, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD has been created

REFERENCES:
- [Derived] Charlson M, Wells M, Devine CM, Watts J, Ramos R, Hollenberg J, Winston G, Phillips E, Wethington E. Interval life events are an important determinant of heterogeneity in outcomes in a randomised trial: a novel, simple method of assessment. BMJ Open. 2024 Jul 30;14(7):e074623. doi: 10.1136/bmjopen-2023-074623. PMID 39079918
- [Derived] Phillips EG, Wells MT, Winston G, Ramos R, Devine CM, Wethington E, Peterson JC, Wansink B, Charlson M. Innovative approaches to weight loss in a high-risk population: The small changes and lasting effects (SCALE) trial. Obesity (Silver Spring). 2017 May;25(5):833-841. doi: 10.1002/oby.21780. Epub 2017 Apr 5. PMID 28382755